CLINICAL TRIAL: NCT06542003
Title: Movin' & Groovin' for Wellness: A Drumming and Dancing Program to Support Well-being in NUS Students
Brief Title: The Impact of Performing Arts on Mental Health, Social Connection, and Creativity in University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Kathleen Rose Agres, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NUS-IRB-2023-3
Record Dates: First submitted 2024-08-03; First posted 2024-08-07 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Mental Health; Quality of Life; Social Isolation; Creativity
Keywords: mental health; social connection; creative expression; arts and health; music intervention; dancing; drumming; performing arts
MeSH Terms: conditions — Psychological Well-Being; Social Isolation; Arts syndrome | interventions — Health

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to two primary groups: an intervention group and a control group. Within the intervention group, participants are further divided into two subgroups due to logistical reasons, allowing for separate sessions for music and dance activities. This division is not to provide different interventions, but rather to manage the logistics of hosting the sessions, e.g. where only so many students may participate in group drumming at a time.
Masking Description: Because participants are either actively receiving facilitated participatory arts sessions or not, it is not possible to mask the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MGW Drum and Dance Group (Experimental): Participants in the intervention group engage in a 10-week program that includes both drumming and dancing sessions. The group is further divided into two subgroups due to logistical reasons, with one subgroup attending five weeks of drumming sessions followed by five weeks of dancing sessions, and the other subgroup attending sessions in the opposite order. All participants in this arm participate in both drumming and dancing sessions.
  Interventions: Behavioral: Movin' and Groovin' for Wellness
- No-treatment Control Group (No Intervention): Participants in the control group do not participate in the drumming and dancing sessions. They represent "normal student life". They only complete the same questionnaires at the same time points as the intervention group to serve as a baseline comparison for evaluating the impact of the interventions.

INTERVENTIONS:
Behavioral: Movin' and Groovin' for Wellness — Movin' and Groovin' for Wellness (MGW) is a 10-week program consisting of facilitated drumming and dancing sessions. The sessions include guided activities involving drumming, dancing, and group improvisation. Each session lasts approximately 1.5 hours, with activities designed to improve mental well-being, enhance social connections, and foster creative expression. The sessions are guided by professional facilitators.
  Arms: MGW Drum and Dance Group

SUMMARY:
The goal of this clinical trial is to investigate whether the "Movin' & Groovin' for Wellness" (MGW) performing arts program is able to support mental, social, and emotional health in NUS students. It will also assess the program's impact on students' well-being. The main questions it aims to answer are:

1. Does participation in the program decrease depressive symptoms, stress levels and anxiety?
2. Does the program foster creative expression among participants?
3. Does the program foster social connections among participants?

Researchers compare the effects of the facilitated music and dance sessions (MGW program) to a Control group that does not participate in these activities. Participants are randomly assigned into either the Experimental (MGW) group or Control group.

Those in the Experimental group are randomly allocated to one of two subgroups, where participants either experience drumming or dancing sessions first (for 5 weeks), followed by the other activity (e.g., the only difference between subgroups is the order in which they experience the facilitated sessions). Both the drumming and dancing sessions are led by trained professionals. The sessions are held weekly for 10 weeks in dedicated performance rooms. Participants also complete questionnaires, and have the opportunity to participate in a focus group discussion to provide feedback about the program.

Control group participants complete the same questionnaires at the same time points without participating in the activities. The program aims to evaluate the effectiveness of music and dance in promoting mental health, social well-being, and creativity among university students.

ELIGIBILITY:
Inclusion Criteria:

* Be currently enrolled in NUS
* Be between the ages of 18-40 years old
* Be fluent (speak and write) in English
* Able to commit to attending the live sessions for the entire 10-week period
* Have normal or corrected-to-normal hearing and vision

Exclusion Criteria:

* Have been diagnosed with a neurological or hearing impairment, or a physical impairment that would prevent moving/dancing
* Are taking medicine to treat their mental health (as this would be a confound in the study)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2023-08-29 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in depressive symptoms, stress levels and anxiety levels | Baseline, Week 5, Week 10
  Measurement of participants' depressive symptoms, stress levels and anxiety levels using the Depression, Anxiety, and Stress Scale (DASS-21). The scores from the DASS-21 questionnaire are used to assess these changes. Depression/Anxiety/Stress sub-scales' scores can range from 0-21 with higher scores indicating worse symptoms.
Changes in quality of life | Baseline, Week 5, Week 10
  Measurement of participants' quality of life using the WHO Quality of Life-BREF (WHOQOL-BREF). This measure captures physical health, psychological health, social relationships, and environmental domains. The physical, psychological, social, and environmental domain scores each range from 4-20 with higher scores indicating a higher quality of life.

SECONDARY OUTCOMES:
Changes in social connection | Baseline, Week 5, Week 10
  Measurement of participants' social networks using the Short Form Lubben Social Network Scale. This scale evaluates the frequency and quality of participants' social interactions. The Friend sub-scale scores range from 0-15 with higher scores indicating more social connection with friends. The Family sub-scale scores range from 0-15 with higher scores indicating greater social connection with family.
Changes in creativity | Baseline, Week 5, Week 10
  Measurement of participants' creative experiences using the Experience of Creation Scale. This scale assesses the impact of creative activities on participants' feelings of empowerment, freedom to decide, impact, and creativity. The scores range from 4-20 with higher scores indicating better experience of creation.
Changes in resilience | Baseline, Week 5, Week 10
  Measurement of emotional resilience using the Brief Resilient Coping Scale. This scale measures participants' ability to cope with stress and adapt to changes, with higher scores indicating better resilience. The scores range from 4-20 with higher scores indicating high resilient copers.
Changes in mood regulation through music | Baseline, Week 5, Week 10
  Measurement of participants' use of music for mood regulation using the Brief Music in Mood Regulation Scale (B-MMR). This scale evaluates various strategies of music listening that individuals use to manage their mood and emotions. For each sub-scale, the scores range from 3-15 with higher scores indicating greater use of that listening strategy for mood regulation.
Participant experience | Week 5, Week 10
  Collection of participants' experience in the program. The bespoken survey asks about students' experiences in the program, spanning artistic engagement, creative expression, comfort, mood, sense of well-being, and social aspects of the program.
Qualitative feedback from focus group discussion | Within two weeks post-program completion
  Collection of lived experience from focus group discussion (FGD) about the program's impact on mental health, social connection, and creativity, as well as general feedback about the MGW program.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen R Agres, PhD, Principal Investigator — National University of Singapore
Locations (1):
- YST Conservatory, 3 Conservatory Drive, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
The IPD won't be shared.

REFERENCES:
- [Derived] Agres KR, Chen Y. The impact of performing arts on mental health, social connection, and creativity in university students: a Randomised Controlled Trial. BMC Public Health. 2025 May 2;25(1):1628. doi: 10.1186/s12889-025-22552-3. PMID 40316963